CLINICAL TRIAL: NCT03332082
Title: A Clinical Trial on the Use of a Commercial Available Tooth Positioner for the Treatment of Simple Orthodontic Relapse
Brief Title: A Commercial Available Tooth Positioner for the Treatment of Simple Orthodontic Relapse
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: losing of funding for the study
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Chung How Kau, Professor and Chair, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300000946
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Orthodontics; Orthodontic Appliance

STUDY DESIGN:
Intervention Model Description: 20 patients will be recruited and treated with a commercially available tooth positioner. The results will be compared with the other group from previously treated patients who were in the alignment phase of Orthodontics.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tooth positioner treatment group (Experimental): The participants that meet the inclusion criteria will be treated with tooth positioner.
  Interventions: Procedure: Tooth positioner

INTERVENTIONS:
Procedure: Tooth positioner — Orthodontic Tooth positioners treatment have been used in the Orthodontic Industry for many years. These positioners are used for small minor movements to complete the final smile. These positioners are made from a biocompatible and FDA approved clear silicone material after the teeth have been set to the final position.

SUMMARY:
Orthodontic relapse occurs in almost 80% of Orthodontic Treatment. The only prevention to phenomenon is the use of fixed retainers or life time active retention. Unfortunately, patients do not comply and after a year of treatment, many stop wearing their retainers and Orthodontic relapse occurs.

The aim of this project is to prospectively analyze the treatment result of consecutive treated patients who have had active orthodontic relapse. 20 patients will be recruited through advertisement to the Department of Orthodontics at the University of Alabama at Birmingham (UAB). The sample will comprise of 20 patients with Class I malocclusions. The records to be collected will comprise of clinical pictures and pre and post study casts. The 3D study casts will be evaluated using the Little's Index. The results will be analyzed with the paired t-test and ANOVA, using the Statistical Analysis System (SAS/STAT®) software.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent dentition
2. Class I malocclusion with crowding or spacing of less than 6 mm for mandibular or maxillary incisors, lower number 1's through 3's
3. Predicted compliance with device use, as determined by the investigator orthodontist
4. Good oral hygiene, as determined by the investigator orthodontist
5. At least average intelligence, as determined by investigator orthodontist

Exclusion Criteria:

1. Any medical or dental condition that in the opinion of the investigator could impact study results during the expected length of the study
2. Patient is currently using any investigational drug or any other investigational device
3. Patient plans to relocate or move within six months of enrollment
4. Allergic to acetaminophen (use of aspirin or non-steroidal anti-inflammatory drugs is excluded for patients while on the study)
5. Use of bisphosphonates, such as osteoporosis drugs, during the study
6. Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The Little's Index | Movement will be recorded by capturing the start and end point of the 6 anterior teeth before and at the completion of the treatment respectively. The duration of the treatment will be up to 10 months.
  The Little's Index of Displacement score will be the primary clinical endpoint used to judge patient success (i.e., effectiveness).

IPD SHARING:
Plan to Share IPD: Undecided